CLINICAL TRIAL: NCT04262869
Title: Phase 2 Study of Platinum-Based Chemotherapy in Combination With Durvalumab (MEDI 4736) for NSCLC in Patients With a Poor Performance Status and the Elderly
Brief Title: Platinum-Based Chemotherapy and Durvalumab for the Treatment of Stage IIIB or IV Non-small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to accrual issues
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Conor Steuer, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00114607; NCI-2019-06508 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4802-19 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2020-02-07; First posted 2020-02-10 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage IIIB Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Carboplatin; durvalumab; Immunoglobulin G; Disulfides; Paclitaxel; Taxes; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (squamous NSCLC) (Experimental): Patients receive carboplatin IV over 15-60 minutes, paclitaxel IV over 3 hours and durvalumab IV over 1 hour on day 1. Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients who do not progress receive durvalumab IV every 4 weeks for up to 35 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Biological: Durvalumab; Drug: Paclitaxel
- Arm II (non-squamous NSCLC) (Experimental): Patients receive carboplatin IV over 15-60 minutes, pemetrexed IV over 10 minutes and durvalumab IV over 1 hour on day 1. Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients who do not progress receive durvalumab IV and pemetrexed IV every 3 weeks for up to 35 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Biological: Durvalumab; Drug: Pemetrexed

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm I (squamous NSCLC)
Drug: Pemetrexed — Given IV
  Other Names: MTA; Multitargeted Antifolate
  Arms: Arm II (non-squamous NSCLC)

SUMMARY:
This phase II trial studies how well platinum-based chemotherapy works when given together with durvalumab in treating patients with stage IIIB or stage IV non-small cell lung cancer. Drugs used in chemotherapy, such as carboplatin, paclitaxel, and pemetrexed, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as durvalumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. The purpose of this study is to find out if the combination of chemotherapy in combination with the immune therapy drug durvalumab would be efficacious and have an acceptable toxicity profile in patients with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the 6-months progression-free survival (PFS) rate with the combination of dose attenuated doublet chemotherapy with durvalumab in advanced non-small cell lung cancer (NSCLC) patients with Eastern Cooperative Oncology Group (ECOG) performance status (PS) 2 status or age >= 70.

SECONDARY OBJECTIVES:

I. To investigate overall response rate. II. To determine the safety profile of the regimen. III. To determine the median PFS and overall survival.

EXPLORATORY OBJECTIVE:

I. Exploratory investigation of biomarkers that could potentially serve as predictive indicators: characterize immunoprofile in peripheral blood by flow cytometry.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I (SQUAMOUS NSCLC): Patients receive carboplatin intravenously (IV) over 15-60 minutes, paclitaxel IV over 3 hours and durvalumab IV over 1 hour on day 1. Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients who do not progress receive durvalumab IV every 4 weeks for up to 35 cycles in the absence of disease progression or unacceptable toxicity.

ARM II (NON-SQUAMOUS NSCLC): Patients receive carboplatin IV over 15-60 minutes, pemetrexed IV over 10 minutes and durvalumab IV over 1 hour on day 1. Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients who do not progress receive durvalumab IV and pemetrexed IV every 3 weeks for up to 35 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol
* Have a histologically confirmed or cytologically confirmed diagnosis of stage IIIB or stage IV NSCLC
* Have a performance status of 2 on the Eastern Cooperative Oncology Group (ECOG) performance status with any age, or age >= 70 with ECOG PS of 0, 1, or 2, on the day of signing informed consent
* Patients must have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as determined by local site investigator/radiology assessment. Target lesions situated in previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* Have not received prior systemic treatment for their advanced/metastatic NSCLC. Subjects who received adjuvant or neoadjuvant therapy are eligible if the adjuvant/neoadjuvant therapy was completed at least 12 months prior to the development of metastatic disease
* Body weight > 30 kg
* Hemoglobin >= 9.0 g/dL
* Absolute neutrophil count (ANC) >= 1.5 (>= 1500 per mm^3)
* Platelet count >= 100) x 10^9/L (>= 100,000 per mm^3)
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN). (This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed if =< 3.0 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be =< 5 x ULN
* Measured creatinine clearance (CL) > 40 mL/min or calculated creatinine CL > 40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976)
* The effects of the study drug on the developing human fetus are unknown. For this reason female of child-bearing potential (FCBP) must have a negative serum or urine pregnancy test prior to starting therapy
* FCBP and men must agree to use adequate contraception (at least one highly effective method and one additional method of birth control at the same time or complete abstinence) prior to study entry, for the duration of study participation and for at least 4 months following study drug discontinuation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. A female of childbearing potential (FCBP) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months (if age > 55 years); if the female subject is < 55 years and she has been naturally postmenopausal for > 1 year her reproductive status has to be verified by additional lab tests (< 20 estradiol OR estradiol < 40 with follicle stimulating hormone [FSH] > 40 in women not on estrogen replacement therapy)
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

* Participation in another clinical study with an investigational product during the last 4 weeks
* ECOG PS 3 or higher
* Prior systemic therapy for the treatment of advanced or metastatic NSCLC
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Completed palliative radiotherapy within 7 days of the first dose of trial treatment
* Has a known sensitivity to any component of carboplatin, pemetrexed, paclitaxel, or durvalumab
* Is unable to unwilling to take folic acid of vitamin b12 supplementation (if non-squamous histology)
* Any unresolved toxicity National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade >= 2 from previous anticancer therapy with the exception of vitiligo, and the laboratory values defined in the inclusion criteria
* Patients with grade >= 2 neuropathy will be evaluated on a case-by-case basis after consultation with the study physician
* Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the study physician
* Any concurrent chemotherapy, investigational product (IP), biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable
* History of allogenic organ transplantation
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events (AEs) or compromise the ability of the patient to give written informed consent
* Prior invasive malignancy (except non-melanomatous skin cancer, low or intermediate risk prostate cancer, or in situ carcinoma fully resected) unless disease free for a minimum of one year
* History of leptomeningeal carcinomatosis
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are clinically stable for at least 2 weeks. Subjects with asymptomatic brain metastases may participate, but will require regular imaging of the brain as a site of disease
* History of active primary immunodeficiency
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis [TB] testing in line with local practice), hepatitis B (known positive hepatitis B virus [HBV] surface antigen [HBsAg] result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for 20. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (hepatitis C virus [HCV]) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA)
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed << 10 mg/day >> of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication)
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
* Patients may not have received prior anti-PD-1, anti PD-L1 including durvalumab or anti CTLA-4 drugs
* Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2021-10-18 (Actual)

PRIMARY OUTCOMES:
6-months progression-free survival (PFS) rate | 6 months
  Will be calculated as proportion along with 95% confidence intervals (CI) using the Clopper-Pearson method. Chi-square test or Fisher's exact test will be used to compare the 6-months PFS rate between the different groups stratified by different factors, respectively. Logistics regression model will be further employed to test the adjusted effect of each factor on 6-month PFS rate after adjusting for other clinical factors and demographic factors.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 5 years
  Will be estimated with the Kaplan-Meier method and compared between different groups using the log-rank test, respectively. The OS of each patient group at specific time points, such as 6 months, 1 year, 3 year, and 5 year, etc. will be also estimated alone with 95% CI. Cox proportional hazards models will be further used in the multivariable analyses to assess adjusted effect of dose levels on the patients' OS after adjusting for other factors. Interaction terms between these factors will also be tested for statistical significance. The proportional hazards assumption will be evaluated graphically and analytically with regression diagnostics. Violations of the proportional hazards assumptions will be addressed by use of time-dependent covariates or extended Cox regression models.
PFS | Up to 5 years
  Will be estimated with the Kaplan-Meier method and compared between different groups using the log-rank test, respectively. The PFS of each patient group at specific time points, such as 6 months, 1 year, 3 year, and 5 year, etc. will be also estimated alone with 95% CI. Cox proportional hazards models will be further used in the multivariable analyses to assess adjusted effect of dose levels on the patients' PFS after adjusting for other factors. Interaction terms between these factors will also be tested for statistical significance. The proportional hazards assumption will be evaluated graphically and analytically with regression diagnostics. Violations of the proportional hazards assumptions will be addressed by use of time-dependent covariates or extended Cox regression models.
Incidence of adverse events (AEs) | Up to 90 days post treatment
  Safety profile of the regimen will be listed and summarized overall and by prognostic factor. Adverse events will also be listed by severity, seriousness, and by system organ class. The number and percentage of subjects who experience AEs will be presented in tabular and/or graphical format and summarized descriptively, where appropriate. No formal statistical comparison between the different factors will be performed. AEs will be presented with and without regard to causality based on the investigator's judgment. The frequency of overall toxicity, categorized by toxicity grades 1 through 5, will be described. Additional summaries will be provided for AEs that are observed with higher frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Conor E Steuer, Principal Investigator — Emory University Hospital/Winship Cancer Institute

IPD SHARING:
Plan to Share IPD: No
Results of the trial and not individual patient data will be shared. The study protocol, consent, and investigator's brochure will be available. The statistical plan is incorporated into the protocol, along with inclusion and exclusion criteria.